CLINICAL TRIAL: NCT04513483
Title: The Effect of Continuous Positive Airway Pressure in Patients With Obstructive Sleep Apnea and Paroxysmal Atrial Fibrillation
Brief Title: CPAP in AF Patients With OSA
Acronym: CPAPAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202002128RINC
Record Dates: First submitted 2020-08-06; First posted 2020-08-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Sleep Apnea
Keywords: Atrial Fibrillation; sleep apnea
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP treatment for 12 months (Experimental): CPAP treatment for 12 months
  Interventions: Device: continuous positive airway pressure
- Placebo (Placebo Comparator): observation
  Interventions: Device: Placebo

INTERVENTIONS:
Device: continuous positive airway pressure — CPAP treatment at night. Treat AF as cardiologist's discretion.
  Arms: CPAP treatment for 12 months
Device: Placebo — Observation. Treat AF as cardiologist's discretion.
  Arms: Placebo

SUMMARY:
Obstructive sleep apnea is associated with atrial fibrillation. This study is to evaluate the effect of continuous positive airway pressure on the burden of atrial fibrillation in the patients with obstructive sleep apnea and paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
Traditional risk factors for AF were established from the original Framingham Heart Study cohort which showed aging, hypertension, congestive heart failure, coronary artery disease, valvular heart disease and diabetes mellitus (DM) as independent risk factors. In the past decade, several important risk factors not encompassed in previous studies have also been found to have a link with AF. One of these newly-identified risk factors is obstructive sleep apnea (OSA), which has been listed as one of the risk factor needed to be assessed and treated in AF patients.

OSA and AF often co-exist and indeed share some risk factors, such as hypertension. AF Patients are more likely to have OSA, with reported prevalence rates of OSA (apnea-hypopnea index [AHI] ≥15) as high as 62% in AF cohorts from hospital-based studies. In community-based cohort studies, a cross-sectional analysis from sleep heart health study (SHSS) found those with sleep-disordered breathing(SDB)/sleep apnea (SA) (respiratory disturbance index [RDI] ≥ 30) had four times the odds of a polysomnography (PSG)-detected nocturnal AF as compared to those without SDB/SA after adjusting confounders. Following from this, a cross-sectional study on Outcomes of Sleep Disorders in Older Men Study (MrOS Sleep Study) showed a dose-response association between RDI and AF.

There are several pathophysiological mechanisms by which OSA could potentially increase the risk of development of new AF, or trigger a recurrence of AF in a patient with an established history of AF. OSA is characterized by repetitive collapse of the upper airway (UA) during sleep. The UA collapses when sleep-related loss in UA dilator muscle tone is superimposed upon a narrow and/or collapsible airway. These obstructive apneas or hypopneas, characterized by unsuccessful inspiratory efforts against an occluded airway, lead to 1) exaggerated negative intrathoracic pressure swings 2) hypoxia, and 3) co-activation of sympathetic and parasympathetic systems, all of which have been shown to potentiate a pro-arrhythmic state. Given that these mechanisms are pro-arrhythmic, CPAP (continuous positive airway pressure), the gold standard therapy for OSA, works by splinting the upper airway open during sleep with subsequent abolition of swings in pressure, hypoxia and arousals, can potentially modify the risk of development of AF or recurrence of AF in OSA patients.

There is a growing body of literature supporting that OSA being as a risk factor for recurrence of AF after cardioversion or ablation and treatment of OSA with CPAP decreased the risk of recurrence of AF. Nevertheless, all of the aforementioned studies are observational or retrospective in nature. Recently, Caples et al. conducted the first randomized control trial using CPAP in patients with AF and OSA but failed to find a difference of recurrence of AF between those treated with CPAP versus usual care. Notably, there are several issues in the study design and methodology that do not allow for firm conclusion from the results of this study. It was a single-center study, enrolling very small number of patients, and used a low cut-off AHI>5/h as inclusion criteria. More importantly, only patients with persistent AF scheduled for cardioversion were included. Given the natural time-course from paroxysmal AF to persistent AF, long-term remodeling or established atrial arrythmogenic substrate in persistent AF may be less or not reversible even when the initial risk factor is removed. In this regard, early intervention with CPAP in patients with paroxysmal AF and OSA, which has never been done in previous studies, should confer a better antiarrythmic effect. Therefore, the investigators aim to test the hypothesis that treatment of OSA with CPAP would reduce the burden of AF in patients with paroxysmal AF.

ELIGIBILITY:
Inclusion Criteria:

1. men or women aged 18 to 80 years
2. paroxysmal AF, diagnosed based on the ACC/AHA/HRS 2014 guideline, and is defined as AF that terminates spontaneously or with intervention within 7 d of onset either by 12-lead EKG, 24-hr Holter, or 14-day ECG monitor.
3. OSA, defined as an AHI>15/hr of sleep, of which >50% of events are obstructive.
4. Informed consent signed

Exclusion Criteria:

1. Moderate-severe valvular heart diseases (regurgitation or stenosis)
2. post heart surgery
3. Uncontrolled systemic hypertension or pulmonary hypertension
4. Use of psychoactive or other drugs that could influence breathing patterns
5. Current use of CPAP treatment
6. Epworth sleepiness scale>10
7. Congestive heart failure (LVEF≦45%)
8. Chronic obstructive pulmonary disease
9. History of stroke or neuromuscular disease
10. Severe insomnia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Change of AF burden | 0, 6, 12 months
  The duration in AF on 14-day ECG monitor (percent)
change of left atrium volume | 0, 6, 12 months
  LA volume index measured by ultrasonocardiography
change of Quality of Life | 0, 6, 12 months
  Questionnaire (Short Form Health Survey-36); higher scores means a better quality of life; maximal score 100%
Number of participants hospitalized for cardiovascular or all causes | 12 months
  Hospitalization for cardiovascular or all causes within the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chieh Yu, MD.PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No